CLINICAL TRIAL: NCT06601829
Title: Congenital Hepatic Fibrosis and Autosomal Recessive Polycystic Kidney Disease in Children at Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sherein Awad Mohamed, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-24-08-01MS
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Congenital Hepatic Fibrosis and Autosomal Recessive Polycystic Kidney Disease in Children at Sohag University Hospital
MeSH Terms: conditions — Hepatic Fibrosis, Congenital

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: abdominal ultrasound — abdominal ulterasound showing multiple cysts in the kidnets and hepatic fibrosis

SUMMARY:
polycystic kidney disease is aherditary disorder characterized by the formation of numerous fluid filled cysts in the kidneys which can lead to progressive renal impairment PKDencompasses aspectrum of disorders with autosomal dominant polycystic kidneydisease and autosomal recessive polycystic kidney disease being the two main types

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged 0-18 years both male and female patients

Exclusion Criteria:

* patients whose guardians dont provide informed consent patients who are not complient with follow up vists and data collection protocols

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cross sectional study prospective and retrospective
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
incidence of congenital hepatic fibrosis in patient with autosomal recessive polycyctic kidney disease | 12 months
  describe congenital hepatic fibrosis in patient with autosomal recessive polycystic kidney explaining their clinical manifestations.diagnosis.managment and complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paul BM, Vanden Heuvel GB. Kidney: polycystic kidney disease. Wiley Interdiscip Rev Dev Biol. 2014 Nov-Dec;3(6):465-87. doi: 10.1002/wdev.152. Epub 2014 Sep 3. PMID 25186187
- [Background] Salman MA, Elgebaly A, Soliman NA. Epidemiology and outcomes of pediatric autosomal recessive polycystic kidney disease in the Middle East and North Africa. Pediatr Nephrol. 2024 Sep;39(9):2569-2578. doi: 10.1007/s00467-024-06281-0. Epub 2024 Jan 23. PMID 38261064
- [Background] Khare A, Krishnappa V, Kumar D, Raina R. Neonatal renal cystic diseases. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2923-2929. doi: 10.1080/14767058.2017.1358263. Epub 2017 Aug 2. PMID 28764564
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Lucchetti L, Chinali M, Emma F, Massella L. Autosomal dominant and autosomal recessive polycystic kidney disease: hypertension and secondary cardiovascular effect in children. Front Mol Biosci. 2023 Mar 10;10:1112727. doi: 10.3389/fmolb.2023.1112727. eCollection 2023. PMID 37006611